CLINICAL TRIAL: NCT04167150
Title: Effect of Montmorency Tart Cherry Supplementation on Bone Biomarkers in Women Aged 65-80 Years: A Pilot Study
Brief Title: Tart Cherry Supplementation and Women's Bone Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oklahoma State University (Other)
Collaborators: Cherry Marketing Institute Research Committee (Unknown)
Responsible Party: Principal Investigator, Brenda Smith, Professor of Nutrition, Oklahoma State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CMI2017-2018
Record Dates: First submitted 2019-11-10; First posted 2019-11-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-11

CONDITIONS: Osteoporosis, Postmenopausal; Osteoporosis, Age-Related
Keywords: osteoporosis; biomarkers; tart cherry; functional food
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis

STUDY DESIGN:
Intervention Model Description: Randomized dose-response pre-test, post-test study design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose 1 (Active Comparator): Participants consume 8 fl oz of tart cherry juice per day.
  Interventions: Dietary Supplement: tart cherry juice concentrate is a commercial product provided by King Orchards (Central Lake, MI)
- Dose 2 (Experimental): Participants consume 2 x 8 fl oz of tart cherry juice per day.
  Interventions: Dietary Supplement: tart cherry juice concentrate is a commercial product provided by King Orchards (Central Lake, MI)

INTERVENTIONS:
Dietary Supplement: tart cherry juice concentrate is a commercial product provided by King Orchards (Central Lake, MI) — Participants were instructed to reconstitute the tart cherry juice concentrate in 8 fl oz of water and consume either 1x or 2x daily for 3 months.

SUMMARY:
In spite of aggressive approaches to prevent and treat osteoporosis, it remains one of the most costly and debilitating diseases associated with aging. The pursuit of alternative approaches for preventing bone loss has included the investigation of a number of promising plant-based foods that can be incorporated into the diet. This project is an extension of our pre-clinical studies with tart cherry, designed to determine whether the findings from our animal study can be extended to humans. Thus, the purpose of this project is to investigate the dose-dependent effect of tart cherry juice consumption on biomarkers of bone metabolism in women, aged 65-80 years. The hypothesis to be tested is that three months of tart cherry supplementation will improve bone biomarkers in a dose-dependent manner. Moreover, these improvements in bone metabolism will correspond to a decrease in markers of inflammation and oxidative stress.

DETAILED DESCRIPTION:
Tart cherries are an excellent course of phenolic compounds and anthocyanins, and in pre-clinical studies have been shown to prevent age-related bone loss. Based on these findings, this pilot study was designed to investigate the effects of three months of tart cherry juice supplementation on improving markers of oxidative stress and bone metabolism in older women. Women (n=30), aged 65-80 yrs, will be recruited for the study and randomly assigned to one of two doses of tart cherry juice (8 or 16 fl oz) per day prepared from a Montmorency cherry concentrate (King Orchards, Central Lake, MI). Study participants will complete two study visits to the Nutritional Sciences Clinical Research Center. At the first visit, informed consent will be obtained and relevant medical history and anthropometric measures will be taken by the research team. A blood draw will be performed to assess baseline, biochemical markers of bone metabolism and inflammation as well as indicators of oxidative status. A physical activity and food frequency questionnaire will be completed by each study participant. Whole body, hip and spine bone density (DXA) scan will be performed by certified bone densitometrist. A 3-month final visit will be scheduled for all study participants in which most of the procedures described at baseline (except DXA) will be repeated. Change in primary and secondary outcome measures (i.e., bone, inflammation and oxidative stress biomarkers) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Women, 65-80 years of age
* Capacity to give informed consent

Exclusion Criteria:

* Hormone replacement therapy in the 3 months prior to starting the study
* Bisphosphonates in the 3 months prior to starting the study
* Raloxifene in the 3 months prior to starting the study
* Intermittent parathyroid hormone in the 3 months prior to starting the study
* Growth hormone or steroids in the 3 months prior to starting the study
* Osteoporosis
* Renal disease
* Cancer
* Cardiovascular disease
* Diabetes
* Respiratory disease
* Gastrointestinal diseases
* Liver disease
* Other chronic conditions that could affect bone metabolism

Ages: 65 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Bone-specific alkaline phosphatase (U/L) | Change from baseline to final visits (3 month intervention)
  Bone formation marker
Tartrate resistant acid phosphatase (U/L) | Change from baseline to final visits (3 month intervention)
  Bone resorption marker

SECONDARY OUTCOMES:
C-reactive protein (mg/L) | Change from baseline to final visits (3 month intervention)
  Marker of inflammation
Thiobarbituric acid reactive species (TBARS) (U/L) | Change from baseline to final visits (3 month intervention)
  Marker of oxidative stress

CONTACTS AND LOCATIONS:
Locations (1):
- Oklahoma State University - Nutritional Sciences, Stillwater, Oklahoma, United States